CLINICAL TRIAL: NCT04143711
Title: A Phase I/II, First-In-Human, Multi-Part, Open-Label, Multiple-Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, Biological, and Clinical Activity of DF1001 in Patients with Locally Advanced or Metastatic Solid Tumors, and Expansion in Selected Indications
Brief Title: Study of DF1001 in Patients with Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dragonfly Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: DF1001-001
Record Dates: First submitted 2019-10-18; First posted 2019-10-29 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Solid Tumor, Adult
Keywords: HER-2; NK Cell; Immunotherapy; Metastatic Breast Cancer; Non-small Cell Lung Cancer; Erbb2; DF1001; Sacituzumab Govitecan-hziy
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Nivolumab; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (22):
- Monotherapy DF1001 Dose Escalation (Experimental): Dose escalation cohorts of DF1001 in sequential ascending order.
  Interventions: Drug: DF1001
- Monotherapy DF1001 Safety/PK/PD Expansion (Experimental): Expansion cohorts of monotherapy DF1001 in multiple dose levels after evaluation for safety in Monotherapy Dose Escalation arm. Additional pharmacokinetic (PK) and pharmacodynamic (PD) samples included in this arm.
  Interventions: Drug: DF1001
- Monotherapy DF1001 Expansion in Urothelial Bladder Cancer (Experimental): Monotherapy expansion cohort enrolling up to 20 patients with urothelial bladder cancer using the recommended phase 2 dose (RP2D) identified in the Monotherapy Dose Escalation arm.
  Interventions: Drug: DF1001
- Monotherapy DF1001 Expansion in Metastatic Breast Cancer (HER2 Low) (Experimental): Monotherapy expansion cohort enrolling up to 20 patients with metastatic breast cancer with documented low expression of HER2 using the recommended phase 2 dose (RP2D) identified in the Monotherapy Dose Escalation arm.
  Interventions: Drug: DF1001
- Monotherapy DF1001 Expansion in Cancers with Erbb2 Amplification (Experimental): Monotherapy expansion cohort enrolling up to 40 patients with solid tumors showing documented erbb2 amplification using the recommended phase 2 dose (RP2D) identified in the Monotherapy Dose Escalation arm.
  Interventions: Drug: DF1001
- Combination Therapy with DF1001 and Nivolumab (Experimental): Combination dose escalation of DF1001 in combination with nivolumab in patients with select solid tumors.
  Interventions: Drug: DF1001; Drug: Nivolumab
- Combination Therapy with DF1001 and Nab-paclitaxel (Experimental): Combination dose escalation of DF1001 in combination with nab-paclitaxel in patients with select solid tumors.
  Interventions: Drug: DF1001; Drug: Nab paclitaxel
- Combination Therapy with DF1001 and Nivolumab Safety/PK/PD Expansion (Experimental): Expansion cohort of DF1001 in combination with nivolumab after evaluation for safety in the Combination Therapy with DF1001 and nivolumab Dose Escalation arm. Additional pharmacokinetic (PK) and pharmacodynamic (PD) samples included in this arm.
  Interventions: Drug: DF1001; Drug: Nivolumab
- Combination Therapy with DF1001 and Nab-paclitaxel Safety/PK/PD Expansion (Experimental): Expansion cohort of DF1001 in combination with nab-paclitaxel after evaluation for safety in the Combination Therapy with DF1001 and nab-paclitaxel Dose Escalation arm. Additional pharmacokinetic (PK) and pharmacodynamic (PD) samples included in this arm.
  Interventions: Drug: DF1001; Drug: Nab paclitaxel
- Combination Therapy with DF1001 and Nivolumab Expansion in Urothelial Bladder Cancer (Experimental): Combination therapy with DF1001 and nivolumab expansion cohort enrolling up to 20 patients with urothelial bladder cancer using the recommended phase 2 dose (RP2D) identified in the Combination Therapy with DF1001 and nivolumab arm.
  Interventions: Drug: DF1001; Drug: Nivolumab
- Monotherapy DF1001 Expansion in Metastatic Breast Cancer (HER2 High) (Experimental): Monotherapy expansion cohort enrolling up to 20 patients with metastatic breast cancer with documented high expression of HER2 using the recommended phase 2 dose (RP2D) identified in the Monotherapy Dose Escalation arm.
  Interventions: Drug: DF1001
- Monotherapy DF1001 Expansion in NSCLC (Experimental): Monotherapy expansion cohort enrolling up to 20 patients with non-small cell lung cancer with documented erbb2 amplification using the recommended phase 2 dose (RP2D) identified in the Monotherapy Dose Escalation arm.
  Interventions: Drug: DF1001
- Combination Therapy with DF1001 and Nivolumab Expansion in NSCLC (Experimental): Combination therapy with DF1001 and nivolumab expansion cohort enrolling up to 20 patients with non-small cell lung cancer with documented low expression of HER2 using the recommended phase 2 dose (RP2D) identified in the Combination Therapy with DF1001 and nivolumab arm.
  Interventions: Drug: DF1001; Drug: Nivolumab
- Monotherapy DF1001 Expansion in Gastric Cancer (Experimental): Monotherapy expansion cohort enrolling up to 20 patients with gastric cancer with documented high expression of HER2 using the recommended phase 2 dose (RP2D) identified in the Monotherapy Dose Escalation arm.
  Interventions: Drug: DF1001
- Combination Therapy with DF1001 and Nivolumab Expansion in Gastric Cancer (Experimental): Combination therapy with DF1001 and nivolumab expansion cohort enrolling up to 20 patients with gastric cancer with documented low expression of HER2 using the recommended phase 2 dose (RP2D) identified in the Combination Therapy with DF1001 and nivolumab arm.
  Interventions: Drug: DF1001; Drug: Nivolumab
- Monotherapy DF1001 Expansion in Esophageal Cancer (Experimental): Monotherapy expansion cohort enrolling up to 20 patients with esophageal cancer with documented high expression of HER2 using the recommended phase 2 dose (RP2D) identified in the Monotherapy Dose Escalation arm.
  Interventions: Drug: DF1001
- Combination Therapy with DF1001 and Nivolumab Expansion in Esophageal Cancer (Experimental): Combination therapy with DF1001 and nivolumab expansion cohort enrolling up to 20 patients with esophageal cancer with documented low expression of HER2 using the recommended phase 2 dose (RP2D) identified in the Combination Therapy with DF1001 and nivolumab arm.
  Interventions: Drug: DF1001; Drug: Nivolumab
- Monotherapy DF1001 Exploratory Efficacy Expansion in NSCLC (Experimental): Monotherapy expansion cohort enrolling up to 20 patients with non-small cell lung cancer with documentation of HER2 activation.
  Interventions: Drug: DF1001
- Combo Therapy with DF1001 and Sacituzumab Govitecan-hziy Exploratory Efficacy Expansion in NSCLC (Experimental): Combination therapy with DF1001 and sacituzumab govitecan-hziy cohort enrolling up to 20 patients, including safety lead-in, with non-small cell lung cancer with documentation of HER2 activation.
  Interventions: Drug: DF1001; Drug: Sacituzumab Govitecan-hziy
- Monotherapy DF1001 Exploratory Efficacy Expansion in Metastatic Breast Cancer (HR+/HER2-) (Experimental): Monotherapy expansion cohort enrolling up to 20 patients with metastatic breast cancer with documentation of HR positive and HER2 negative expression.
  Interventions: Drug: DF1001
- DF1001 with Sacituzumab Govitecan-hziy Exploratory Efficacy Expansion in Breast Cancer (HER2+) (Experimental): Combination therapy with DF1001 and sacituzumab govitecan-hziy cohort enrolling up to 40 patients, including safety lead-in, with metastatic breast cancer with documentation of HER2 positive expression.
  Interventions: Drug: DF1001; Drug: Sacituzumab Govitecan-hziy
- DF1001 with Sacituzumab Govitecan-hziy Exploratory Efficacy Expansion in Breast Cancer (HR+/HER2-) (Experimental): Combination therapy with DF1001 and sacituzumab govitecan-hziy cohort enrolling up to 40 patients, including safety lead-in, with metastatic breast cancer with documentation of HR positive and HER2 negative expression.
  Interventions: Drug: DF1001; Drug: Sacituzumab Govitecan-hziy

INTERVENTIONS:
Drug: DF1001 — Immunotherapy agent targeting NK cells.
Drug: Nivolumab — Anti-PD-1 immunotherapy agent
  Arms: Combination Therapy with DF1001 and Nivolumab; Combination Therapy with DF1001 and Nivolumab Expansion in Esophageal Cancer; Combination Therapy with DF1001 and Nivolumab Expansion in Gastric Cancer; Combination Therapy with DF1001 and Nivolumab Expansion in NSCLC; Combination Therapy with DF1001 and Nivolumab Expansion in Urothelial Bladder Cancer; Combination Therapy with DF1001 and Nivolumab Safety/PK/PD Expansion
Drug: Nab paclitaxel — A chemotherapy treatment combining paclitaxel with albumin
  Arms: Combination Therapy with DF1001 and Nab-paclitaxel; Combination Therapy with DF1001 and Nab-paclitaxel Safety/PK/PD Expansion
Drug: Sacituzumab Govitecan-hziy — A Trop-2 (Tumor-associated calcium signal transducer 2) directed antibody and topoisomerase inhibitor drug conjugate
  Arms: Combo Therapy with DF1001 and Sacituzumab Govitecan-hziy Exploratory Efficacy Expansion in NSCLC; DF1001 with Sacituzumab Govitecan-hziy Exploratory Efficacy Expansion in Breast Cancer (HER2+); DF1001 with Sacituzumab Govitecan-hziy Exploratory Efficacy Expansion in Breast Cancer (HR+/HER2-)

SUMMARY:
DF1001-001 is a study of a new molecule that targets natural killer (NK) cells and T-cell activation signals to specific receptors on cancer cells. The study will occur in two phases. The first phase will be a dose escalation phase, enrolling patients with various types of solid tumors that express human epidermal growth factor receptor 2 (HER2). The second phase will include a dose expansion using the best dose selected from the first phase of the study. Multiple cohorts will be opened with eligible patients having either HER2 activated non-small cell lung cancer, hormone receptor (HR) positive HER2 negative metastatic breast cancer, or HER2 positive metastatic breast cancer. DF1001-001 will be administered as monotherapy or in combination; combinations are DF1001 + nivolumab, DF1001 + Nab paclitaxel, and DF1001 + sacituzumab govitecan-hziy.

ELIGIBILITY:
Inclusion Criteria: General (applies to all cohorts)

1. Signed written informed consent.
2. Male or female patients aged ≥ 18 years.
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at study entry and an estimated life expectancy of at least 3 months.
4. Baseline Left Ventricular Ejection Fraction (LVEF) ≥ 55% measured by echocardiography (preferred) or multigated acquisition (MUGA) scan.
5. Adequate hematological function.
6. Adequate hepatic function.
7. Adequate renal function.
8. Effective contraception for women of child bearing potential (WOCBP) patients as defined by World Health Organization (WHO) guidelines for 1 "highly effective" method or 2 "effective" methods.

Inclusion Criteria: NSCLC (HER2 Activated) Exploratory Efficacy Cohorts - Monotherapy and Combination with Sacituzumab Govitecan-hziy.

1. Have progression of unresectable locally advanced or metastatic NSCLC after last systemic therapy (as confirmed by investigator) or be intolerant of last systemic therapy.
2. Have HER2 overexpression status (IHC 2+ or 3+), or ERBB2 amplification, or HER2 activating mutation
3. Have recurrent or progressive disease during or after platinum doublet-based chemotherapy.
4. Have received and progressed on or after anti-PD-(L)1 therapy.

Inclusion Criteria: Metastatic Breast Cancer (HR+/HER2-) Exploratory Efficacy Cohort - Monotherapy and Combination with Sacituzumab Govitecan-hziy.

1. Documented evidence of HR+ metastatic breast cancer
2. Documented evidence of HER2- status.
3. Disease progression or recurrence after prior therapy.

Inclusion Criteria: Metastatic Breast Cancer (HER2+) Exploratory Efficacy Cohorts - Combination with Sacituzumab Govitecan-hziy

1. Have histologically confirmed HER2+ breast cancer.
2. Have received prior treatment with trastuzumab, pertuzumab, ado-trastuzumab emtansine (T-DM1), or trastuzumab deruxtecan (T-DXd).
3. Have progression of unresectable locally advanced metastatic breast cancer after last systemic therapy or be intolerant of last systemic therapy.

Inclusion Criteria: Dose Escalation

1. Evidence of objective disease, but participation does not require a measurable lesion.
2. Locally advanced or metastatic solid tumors, for which no standard therapy exists, or standard therapy has failed.
3. HER2 expression by immunohistochemistry and/or erbb2 amplification and/or erbb2 activating mutations.

Inclusion Criteria: "3+3" Nivolumab Combination Cohort

1. Eligible to receive nivolumab per its label for a malignancy of epithelial origin; or
2. Have no standard therapy available, or standard therapy has failed, and must not have received nivolumab prior to joining the study.
3. HER2 expression by immunohistochemistry and/or ebb2 amplification and/or erbb2 activating mutations must be documented on either archival tissue or fresh tumor biopsy.

Inclusion Criteria: "3+3" Nab paclitaxel Combination Cohort

1. Patients must be eligible for treatment with nab-paclitaxel per its label, or have no standard therapy available, or standard therapy has failed.
2. HER2 expression by immunohistochemistry and/or erbb2 amplification and/or erbb2 activating mutations must be documented on either archival tissue or fresh tumor biopsy.

Inclusion Criteria: Safety/PK/PD Expansion Cohorts (Monotherapy and Combination Therapy).

1. Fresh tumor biopsy must be obtained during the screening window.
2. HER2 expression by immunohistochemistry (IHC).
3. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.

Inclusion Criteria: Urothelial Bladder Cancer Expansion Cohort(s).

1. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
2. Histologically or cytologically documented locally advanced or metastatic transitional cell carcinoma of the urothelium (including renal pelvis, ureters, urinary urothelial, urethra).
3. Patients must have received a platinum containing chemotherapy and an anti PD-1 or anti PD-L1 for the treatment of urothelial bladder cancer.

Inclusion Criteria: Breast Cancer (HER2 Low) Expansion Cohort

1. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1
2. Histologically documented (metastatic or locally advanced) breast cancer.
3. Absence of erbb2 amplification by ISH and/or HER2 IHC of 0, 1+, or 2+.
4. Patient must have progressed after one line of systemic chemotherapy.

Inclusion Criteria: Breast Cancer (HER2 High) Expansion Cohort

1. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1
2. Histologically documented (metastatic or locally advanced) breast cancer.
3. Erbb2 amplification by ISH and/or HER2 IHC of 3+, or 2+. If Herceptest score is 2+, ISH results should demonstrate erbb2 amplification.

Inclusion Criteria: Basket erbb2 amplified Expansion Cohort

1. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
2. Documented history of erbb2 amplification.
3. Patients must have received at least one line of an approved or established therapy.

Inclusion Criteria: Gastric Cancer (HER2 High) Expansion Cohort

1. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
2. Advanced (unresectable/recurrent/metastatic) gastric cancer or cancer of the gastro-esophageal junction.
3. Tumor must have been declared HER2 positive.

Inclusion Criteria: Gastric Cancer (HER2 Low) Expansion Cohort

1. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
2. Advanced (unresectable/recurrent/metastatic) gastric cancer or cancer of the gastro-esophageal junction.
3. Tumor must have been declared HER2 low; ISH non-amplified and/or HER2 IHC of 0, 1+ or 2+. If Herceptest score is 0, HER2 must be detected by IHC on at least 1+ of the tumor cells.

Inclusion Criteria: Esophageal Cancer (HER2 High) Expansion Cohort

1. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
2. Advanced (unresectable/recurrent/metastatic) esophageal cancer.
3. Tumor must have been declared HER2 positive.

Inclusion Criteria: Esophageal Cancer (HER2 Low) Expansion Cohort

1. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
2. Advanced (unresectable/recurrent/metastatic) esophageal cancer.
3. Tumor must have been declared HER2 low; ISH non-amplified and/or HER2 IHC of 0, 1+ or 2+. If Herceptest score is 0, HER2 must be detected by IHC on at least 1+ of the tumor cells.

Inclusion Criteria: Non-small Cell Lung Cancer (HER2 Low) Expansion Cohort

1. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
2. Histologically confirmed NSCLC meeting stage criteria for stage IIIB, stage IV, or recurrent disease that has been confirmed to have HER2 expression (at least 1+, however, patients must not carry an erbb2 amplification) via archival or fresh biopsy tissue prior to study enrollment.
3. Patients must have recurrent or progressive disease during or after platinum doublet-based chemotherapy.

Inclusion Criteria: Non-small Cell Lung Cancer (HER2 High) Expansion Cohort

1. Disease must be measurable with at least 1 unidimensional measurable lesion by RECIST 1.1.
2. Histologically confirmed NSCLC meeting stage criteria for stage IIIB, stage IV, or recurrent disease that has been confirmed to have amplification of erbb2 via archival or fresh biopsy tissue prior to study enrollment.
3. Patients must have recurrent or progressive disease during or after platinum doublet-based chemotherapy.

Exclusion Criteria:

1. Concurrent anticancer treatment (eg, cytoreductive therapy, radiotherapy [with the exception of palliative bone directed radiotherapy], immune therapy, or cytokine therapy except for erythropoietin), major surgery (excluding prior diagnostic biopsy), concurrent systemic therapy with steroids or other immunosuppressive agents, or use of any investigational drug within 28 days or 5 half-lives before the start of study treatment. Note: Patients receiving bisphosphonates are eligible provided treatment was initiated at least 14 days before the first dose of DF1001.
2. Previous malignant disease other than the target malignancy to be investigated in this study within the last 3 years, with the exception of basal or squamous cell carcinoma of the skin or cervical carcinoma in situ.
3. Rapidly progressive disease.
4. Active or history of central nervous system (CNS) metastases.
5. Receipt of any organ transplantation including autologous or allogeneic stem-cell transplantation.
6. Significant acute or chronic infections (including historic positive test for human immunodeficiency virus [HIV], or active or latent hepatitis B or active hepatitis C tested during the screening window).
7. Preexisting autoimmune disease (except for patients with vitiligo) needing treatment with systemic immunosuppressive agents for more than 28 days within the last 3 years or clinically relevant immunodeficiencies (eg, dys-gammaglobulinemia or congenital immunodeficiencies), or fever within 7 days of Day 1.
8. Known severe hypersensitivity reactions to mAbs (≥ Grade 3 NCI-CTCAE v5.0), any history of anaphylaxis, or uncontrolled asthma (ie, 3 or more features of partly controlled asthma).
9. Persisting toxicity related to prior therapy > Grade 1 NCI-CTCAE v5.0, however alopecia and sensory neuropathy ≤ Grade 2 is acceptable.
10. Pregnancy or lactation in females during the study.
11. Known alcohol or drug abuse.
12. Serious cardiac illness
13. NYHA III of IV heart failure or systolic dysfunction (LVEF < 55%)
14. High-risk uncontrolled arrhythmias ie, tachycardia with a heart rate > 100/min at rest
15. Significant ventricular arrhythmia (ventricular tachycardia) or higher-grade Atrioventricular block (AV-block; second-degree AV-block Type 2 [Mobitz 2] or third-degree AV-block)
16. Angina pectoris requiring anti-anginal medication
17. Clinically significant valvular heart disease
18. Evidence of transmural infarction on ECG
19. Poorly controlled hypertension (defined by: systolic > 180 mm Hg or diastolic > 100 mm Hg)
20. Clinically relevant uncontrolled cardiac risk factors, clinically relevant pulmonary disease or any clinically relevant medical condition in the opinion of the Investigator that may limit participation in this study.
21. Severe dyspnea at rest due to complications of advanced malignancy or requiring supplementary oxygen therapy.
22. All other significant diseases (e.g., inflammatory bowel disease), which, in the opinion of the Investigator, might impair the patient's ability to participate
23. Any psychiatric condition that would prohibit the understanding or rendering of informed consent.
24. Legal incapacity or limited legal capacity.
25. Incapable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Estimated)
Dates: Start 2019-11-11 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Assessment of number of dose limiting toxicities experienced on study as defined per criteria in the study protocol | First 3 weeks of treatment for each subject.
  To assess the number of adverse events experienced during the study that meet dose limiting toxicity criteria per the study protocol.
Assess Overall Response Rate | Through 90 days after completion of the study, an average of 1 year.
  To assess the confirmed Overall Response Rate (ORR) per RECIST version 1.1 criteria by Investigator Assessment in the Efficacy Phase.
Assess number of adverse events observed during treatment with DF1001 in combination with Nivolumab | Screening visit up to 28 days after last treatment on study.
  To assess the safety of DF1001 in Combination therapy with nivolumab by measuring Number of subjects with Treatment-Emergent Adverse Events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Assess number of adverse events observed during treatment with DF1001 in combination with Nab paclitaxel | Screening visit up to 28 days after last treatment on study.
  To assess the safety of DF1001 in Combination therapy with Nab paclitaxel by measuring Number of subjects with Treatment-Emergent Adverse Events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Assess number of adverse events observed during treatment with DF1001 in combination with Sacituzumab govitecan-hziy | Screening visit up to 28 days after last treatment on study.
  To assess the safety of DF1001 in Combination therapy with Sacituzumab govitecan-hziy by measuring Number of subjects with Treatment-Emergent Adverse Events according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0

SECONDARY OUTCOMES:
Evaluation of DF1001 Pharmacokinetics | From start of treatment up through 28 days after last treatment.
  Concentration vs time of DF1001 will be measured using blood samples taken a various time points on study
Evaluation of DF1001 Immunogenicity | Every 3 weeks up to 28 days after last treatment.
  Evaluate the immunogenicity of DF1001 by measuring the number of patients developing anti-DF1001 antibodies
Assess Overall Survival (OS) Time. | Time from enrollment in the study until death, measured up to 2 years after last treatment on study.
  To assess Overall Survival (OS)
Assess Overall Response Rate by Investigator Assessment. | From time of initiation of therapy until the date of first documented tumor progression, assessed up to 24 months
  To assess confirmed and unconfirmed Overall Response Rate (ORR) by Investigator Assessment for patients enrolled in the dose escalation phase.
Assess Duration of Response by Investigator Assessment. | From time of initiation of therapy until the date of first documented tumor progression, assessed up to 24 months
  To assess Duration of Response (DOR) for confirmed responses by Investigator Assessment for patients enrolled in the dose escalation phase and in the efficacy expansion phase.
Assess Best Overall Response by Investigator Assessment. | Through 90 days after completion of the study, an average of 1 year.
  To assess confirmed Best Overall Response by Investigator Assessment for patients enrolled in the dose escalation phase and in the efficacy expansion phase.
Assess Progression-free Survival by Investigator Assessment. | From time of initiation of therapy until the date of first documented tumor progression, assessed up to 24 months
  To assess Progression-free Survival (PFS) by Investigator Assessment for patients enrolled in the dose escalation phase and in the efficacy expansion phase.

CONTACTS AND LOCATIONS:
Locations (52):
- United States (19):
  - University of California Irvine Medical Center, Irvine, California
  - University of Southern California, Los Angeles, California
  - Sharp Healthcare, San Diego, California
  - University of California San Francisco, San Francisco, California
  - University of Kansas Medical Center Research Institute, Inc., Westwood, Kansas
  - Louisiana State University, New Orleans, Louisiana
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Icahn School of Medicine: Tisch Cancer Institute at Mount Sinai Medical Center, New York, New York
  - Montefiore Einstein Center for Cancer Care, The Bronx, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Abramson Cancer Center, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - MD Anderson Cancer Center, Houston, Texas
  - Multicare Health System Tacoma General Hospital, Tacoma, Washington
  - University of Wisconsin, Madison, Wisconsin
- Belgium (3):
  - Centre Hospitalier de l'Ardenne, Arlon
  - Grand Hopital de Charleroi, Charleroi
  - Domaine Universitaire du Sart Tilman; CHU de Liege, Liège
- Denmark (2):
  - Rigshospitalet, Copenhagen, Capital Region
  - Herlev og Gentofte Hospital, Herlev
- France (11):
  - Institut Curie, Paris, Paris
  - Groupe Hospitalier Saint Andre, Bordeaux
  - Centre Georges-Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Regional du Cancer de Montepelier, Montpellier
  - Groupe Hospitalier Pitie Salpetriere, Paris
  - CHU de Rennes Hopital Pontechaillou, Rennes
  - ICO - Site Rene Gauducheau, Saint-Herblain
  - Institut Claudius Regaud, Toulouse
- Netherlands (6):
  - Amsterdam University Medical Center, Amsterdam
  - Universitair Medisch Centrum Groningen, Groningen
  - Maasticht University Medical Center, Maastricht
  - Radboud University Nijmegen, Nijmegen
  - Erasmus University Medical Center, Rotterdam
  - UMC Utrecht, Utrecht
- South Korea (11):
  - Inje University Haeundae Paik Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - National Cancer Center, Goyang-si
  - Ajou University Hospital, Gyeonggi-do
  - CHA Bundang Medical Center, CHA University, Gyeonggi-do
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Korea University Guro Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul